CLINICAL TRIAL: NCT06977815
Title: Ensayo Clínico No Aleatorizado Sobre la Estimulación Cognitiva Con Realidad Virtual en Pacientes Con Deterioro Cognitivo Leve
Brief Title: Non-randomized Clinical Trial on Cognitive Stimulation With Virtual Reality in Patients With Mild Cognitive Impairment
Acronym: RVEC-DCL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Badalona Serveis Assistencials (Other)
Responsible Party: Principal Investigator, Jose Ferrer Costa, Medical Researcher and Project Manager, Badalona Serveis Assistencials
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PI-24-210
Record Dates: First submitted 2025-05-01; First posted 2025-05-18 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Mild Cognitive Impairment; Cognitive Dysfunction; Aging
Keywords: Virtual Reality; Cognitive Rehabilitation; Older Adults; VR-Enhanced Therapy; Neurocognitive Disorders; Cognitive Stimulation; Gerontology
MeSH Terms: conditions — Cognitive Dysfunction; Neurocognitive Disorders

STUDY DESIGN:
Intervention Model Description: Two groups: one receiving computer-based cognitive rehabilitation with added virtual reality (VR); the other receiving computer-based cognitive rehabilitation only.
Masking Description: No masking; participants and facilitators are aware of group allocation due to the nature of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR-Enhanced Cognitive Rehabilitation (Experimental): Participants receive a computer-based cognitive rehabilitation program supplemented with immersive virtual reality exercises. The program is delivered in two sessions per week over 12 weeks, for a total of approximately 20 to 22 sessions.
  Interventions: Behavioral: VR-Enhanced Cognitive Rehabilitation
- Standard Cognitive Rehabilitation (Active Comparator): Participants receive a standard computer-based cognitive rehabilitation program. The program is delivered in two sessions per week over 12 weeks, for a total of approximately 20 to 22 sessions.
  Interventions: Behavioral: Standard Cognitive Rehabilitation

INTERVENTIONS:
Behavioral: VR-Enhanced Cognitive Rehabilitation — A program consisting of 45-minute computer-based cognitive rehabilitation exercises, enhanced with 15-20 minutes of immersive virtual reality (VR) content per session. The VR component targets memory, attention, and executive function. Sessions are delivered twice per week over 12 weeks.
  Other Names: Virtual Reality Cognitive Support
  Arms: VR-Enhanced Cognitive Rehabilitation
Behavioral: Standard Cognitive Rehabilitation — A program consisting of 45-minute computer-based cognitive rehabilitation exercises targeting memory, attention, and executive function. Sessions are delivered twice per week over 12 weeks. No VR content is included.
  Other Names: Computer-Based Cognitive Training
  Arms: Standard Cognitive Rehabilitation

SUMMARY:
The purpose of this study is to find out if adding virtual reality (VR) to a cognitive training program helps improve cognitive performance in older adults with mild cognitive impairment (MCI). In this study, all participants will take part in a 12-week computer-based cognitive rehabilitation program. One group will also use immersive VR for 15-20 minutes at the end of each session. Participants will attend 2 sessions per week, completing at least 20 sessions and up to 22, depending on the clinic's schedule. Researchers will measure changes in attention, memory, and thinking skills using standard cognitive tests. They will also collect feedback on how participants experience the VR exercises.

DETAILED DESCRIPTION:
This clinical trial evaluates a cognitive rehabilitation program enhanced with virtual reality (VR) for older adults with mild cognitive impairment (MCI). The study investigates whether adding immersive VR exercises to a conventional program improves cognitive performance compared to standard cognitive rehabilitation alone.

All participants take part in a structured, computer-based cognitive training program delivered over 12 weeks. Sessions occur twice per week, with participants completing at least 20 and up to 22 sessions depending on clinic scheduling. The intervention group receives an additional 15-20 minutes of immersive VR content at the end of each session. VR exercises target attention, memory, and executive functioning, aiming to increase engagement and therapeutic value.

This trial complements a previously registered pilot study (ClinicalTrials.gov Identifier: NCT06155721) and builds on its published results.

Cognitive performance will be assessed using standardized neuropsychological tests including the Montreal Cognitive Assessment (MoCA), Mini-Mental State Examination (MMSE), Digit Span, Trail Making Test (TMT), and Symbol Digit Modalities Test (SDMT). Functional capacity will be evaluated using the Lawton-Brody scale. Usability and satisfaction with the VR system will be measured in the intervention group using the System Usability Scale (SUS) and a custom satisfaction questionnaire.

The study has been approved by the Germans Trias i Pujol University Hospital Research Ethics Committee (PI-24-210) and complies with the Declaration of Helsinki and the European General Data Protection Regulation (GDPR).

ELIGIBILITY:
Inclusion Criteria:

* Age between 60 or older
* Clinical diagnosis of mild cognitive impairment (MCI)
* Preserved autonomy in basic and instrumental activities of daily living
* MoCA score between 18 and 26
* Ability to use a computer interface with or without assistance
* Capacity to understand and sign informed consent

Exclusion Criteria:

* Diagnosis of dementia (MMSE < 18 or clinical judgment)
* Severe visual or hearing impairment affecting task participation
* History of epilepsy, vertigo, or conditions contraindicating VR use
* Severe psychiatric or neurological illness (e.g., major depression, Parkinson's disease)
* Enrollment in other cognitive training programs during the study period

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-04 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Global Cognition as Measured by the Montreal Cognitive Assessment (MoCA) | Baseline and immediately post-intervention (Week 12, within 1 week after last session)
  MoCA is a 30-point screening tool for global cognitive function, assessing memory, attention, language, visuospatial skills, and executive function.
  Score Range: 0 to 30 points
  - Higher scores means better global cognition function
Global Cognition as Measured by the Mini-Mental State Examination (MMSE) | Baseline and immediately post-intervention (Week 12, within 1 week after last session)
  MMSE is a 30-point questionnaire evaluating orientation, attention, recall, language, and visual construction Score Range: 0 to 30 points. Higher scores means better global cognition function
Short-Term Memory as Measured by the Digit Span Test (Forward Span) | Baseline and immediately post-intervention (Week 12, within 1 week after last session)
  Forward Digit Span measures verbal short-term memory. Score Range: 0 to 9 points Higher scores reflect better performance.
Working Memory as Measured by the Digit Span Test (Backward Span) | Baseline and immediately post-intervention (Week 12, within 1 week after last session)
  Backward Digit Span assesses working memory and mental manipulation. Score Range: 0 to 9 points. Higher scores indicate better working memory.
Visuospatial Attention as Measured by the Trail Making Test Part A (TMT-A) | Baseline and immediately post-intervention (Week 12, within 1 week after last session)
  TMT-A measures visual attention and processing speed. The outcome is time to completion measured in seconds, typically ranging from several seconds to several minutes.
  Lower times (faster completion) indicate better visuospatial attention.
Executive Function as Measured by the Trail Making Test Part B (TMT-B) | Baseline and immediately post-intervention (Week 12, within 1 week after last session)
  TMT-B assesses alternating attention and executive control. The outcome is time to completion measured in seconds, typically ranging from several seconds to several minutes.
  Lower times (faster completion) indicate better alternating attention.
Processing Speed as Measured by the Symbol Digit Modalities Test (SDMT) | Baseline and immediately post-intervention (Week 12, within 1 week after last session)
  SDMT: Symbol Digit Modalities Test. The Symbol Digit Modalities Test (SDMT) measures processing speed, attention, and visual-motor coordination. During the test, participants are required to match abstract symbols with corresponding numbers using a key. The total raw score is calculated as the number of correct symbol-digit pairs completed within a 90-second interval. There is no fixed maximum score, as it varies based on individual performance.
  Higher scores indicate better processing speed and cognitive performance.
Functional Capacity as Measured by the Lawton-Brody Instrumental Activities of Daily Living Scale | Baseline and immediately post-intervention (Week 12, within 1 week after last session)
  The Lawton-Brody Instrumental Activities of Daily Living Scale evaluates functional independence in activities such as telephone use, shopping, cooking, and managing finances. Scores range from 0 to 8, with higher scores indicating greater independence. Each task is scored as independent (1) or dependent (0).

SECONDARY OUTCOMES:
Patient Usability of the VR System as Measured by the Adapted 8-Item System Usability Scale (SUS) | Post-intervention (Week 12, within 1 week after last session)
  Participants rate the comfort and tolerability of the Meta Quest 2 or 3 headset after the final session. The scale includes 8 items addressing physical discomfort (e.g., weight, visual strain, dizziness, fatigue, and headache).
  Score Range: 0 to 100 (converted from Likert responses) Interpretation: Higher scores indicate greater headset tolerability and comfort.
Patient Comfort and Tolerability of the VR Headset as Measured by an 8-Item Adapted Scale | Post-intervention (Week 12, within 1 week after last session)
  Participants rate the comfort and tolerability of the Meta Quest 2 or 3 headset after the final session. The scale includes 8 items addressing physical discomfort (e.g., weight, visual strain, dizziness, fatigue, and headache).
  Score Range: 0 to 100 (converted from Likert responses) Interpretation: Higher scores indicate greater headset tolerability and comfort.
Clinician Usability of the VR System as Measured by the Adapted 8-Item System Usability Scale (SUS) | Post-intervention (Week 12, within 1 week after last session)
  An adapted SUS completed by professionals delivering the intervention. The 8 items assess perceived usability, integration into clinical workflow, and ease of use for patients.
  Score Range: 0 to 100 Interpretation: Higher scores indicate better usability.
Clinician Perception of VR Headset Comfort for Patients as Measured by a 3-Item Questionnaire | Post-intervention (Week 12, within 1 week after last session)
  Professionals rate their perception of how comfortable and manageable the VR headset is for patients. The 3 items assess concerns such as weight, usability of controls, and prolonged wear tolerance.
  Score Range: 0 to 100 (converted from Likert responses) Interpretation: Higher scores indicate better perceived comfort and usability for patients.

OTHER OUTCOMES:
Participant Age | Baseline
  Age in years, collected at baseline. Used to describe the study population and for subgroup analysis if needed.
Participant Sex | Baseline
  Self-reported biological sex, categorized as:
  0 = Female
  1 = Male 3 = Other Collected at baseline to describe participant characteristics.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Socio Sanitario El Carmen, Badalona, Barcelona, Spain

REFERENCES:
- [Background] Virtual Reality in Cognitive Rehabilitation: A Pilot Study on Usability and Preliminary Clinical Outcomes in Seniors with Mild Cognitive Impairment Jose Ferrer Costa, Maria Jose Ciudad, Maribel González Abad, and José Luis Rodríguez García Journal of Medical Extended Reality 2025 2:1, 30-42